CLINICAL TRIAL: NCT02196246
Title: A Clinical Study to Evaluate the Ability of an iPad Based Photographic Image Analysis System to Discriminate Benign Skin Lesions From Those Considered Suspect for Melanoma
Brief Title: Moletest Clinical Study in Scotland
Status: Completed | Type: Observational
Sponsor: Moletest Scotland Ltd (Industry)
Collaborators: Digital Health & Care Institute (Other); NHS Lanarkshire (Other Government)
Responsible Party: Principal Investigator, Girish Gupta, Principal Investigator Scientic Advisory Board member, Moletest Scotland Ltd
Other Study IDs: Protocol-004
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample of suspect lesion taken for Biopsy, sample is only retained from initial inspection until Biopsy, not other Biospecimen retention is required
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate an iPad based photoimage analysis system (Moletest) for improving discrimination of benign from malignant suspicious skin lesions or moles. Specifically the objective is to demonstrate that the Moletest system is able with a sufficient degree of confidence (95%) to identify lesions which are benign

ELIGIBILITY:
Inclusion Criteria:

All patients referred to the Dermatology Department, Lanarkshire Hospitals during a period to be defined for assessment of suspicious skin lesions (cutaneous moles) will be eligible for inclusion in the study. There are no age limits but patients under the age of 18 years will also have their inclusion subject to parental/guardian consent

Exclusion Criteria:

There is no exclsion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to the Dermatology Department, Lanarkshire Hospitals for assessment of suspicious skin lesions are eligible for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical accuracy of Moletest application, the combined measured attributes of a suspect legion compared to the outcome of a biopsy performed on the legion | 6 weeks turnaround for each sample
  The image and analysis by the application are performed within 10 minutes of the patient giving consent to be part of this study. The biopsy that will be used for comarison with the image analysis will be available to the Investigators approximatly 6 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Peter Freedman, Study Director — Royal College of Physicians
Locations (1):
- NHS Lanarkshire R&D, Airdrie, United Kingdom